CLINICAL TRIAL: NCT05699148
Title: Gut Imaging for Function and Transit in Cystic Fibrosis 3 Junior: an Evaluation of Triple Combination Therapy in Children Aged 6 to 11 Years
Brief Title: Gut Imaging for Function and Transit in Cystic Fibrosis 3 Junior
Acronym: GIFT-CFJunior
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20CS036 sub-study
Record Dates: First submitted 2023-01-10; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CFTR modulators; Gastrointestinal; Lung; Liver; Magnetic resonance imaging; Elexacaftor/ tezacaftor/ ivacaftor
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Children with cystic fibrosis aged 6 to 11 years: Group of children who have at least one copy of Phe508del gene mutation and are eligible for starting on the modulator elexacaftor/ tezacaftor/ ivacaftor (ETI). This group will have baseline MRI scans before starting ETI and aiming to have subsequent scans post starting ETI (6 months to 1 year post starting ETI)
  Interventions: Drug: Elexacaftor / Ivacaftor / Tezacaftor
- Control Group: Age and gender matched controls with no history of cystic fibrosis or gastrointestinal disease. This group will undergo one set of scans only.

INTERVENTIONS:
Drug: Elexacaftor / Ivacaftor / Tezacaftor — Triple combination therapy is licensed in the UK for prescription to paediatric patients aged 6 to 11 years. ETI will be started as part of routine clinical care.
  Other Names: Kaftrio, Trikafta
  Groups: Children with cystic fibrosis aged 6 to 11 years

SUMMARY:
Recently trial data has shown that the medicine KaftrioTM (Elexacaftor/ Tezacaftor/ Ivacaftor) improves lung function in children aged 6 to 11 years who have cystic fibrosis (CF). This has led to it being licensed for use in the UK in 2022 and is now being prescribed in this age group. There is little information in trials however that shows the effect KaftrioTM (ETI) has on the gut or liver in this age group.

Previous studies in the GIFT-CF series (NCT 03566550, NCT04006873 and NCT04618185) has found differences in the functioning of the gut between adults with CF and healthy controls but it is not known whether these differences are present in those aged 6 to 11 years.

This study is a significant amendment of the GIFT-CF3 protocol (NCT04618185) that aims to measure gut function using magnetic resonance imaging (MRI) in children with CF before and after starting ETI. This study also aims to opportunistically measure lung function and structure using MRI and explore how the liver can be measured using MRI in this age group.

The study is split into 2 stages. The first is a pilot stage using the modified GIFT-CF protocol recruiting 3 children with CF before starting ETI and 3 healthy volunteers. This is to determine we are able to successfully perform these scans in these age groups. If successful, the second stage will recruit a further 12 children with CF before they start ETI. This will take our cohort up to 15 children with CF. This cohort will then be rescanned 6 months after starting ETI using the same scan protocol.

DETAILED DESCRIPTION:
This is an observational cohort study using MRI to measure gastrointestinal (GI) function, lung structure and function and liver endpoints in children with CF aged 6 to 11 years. The study will use a modified version of the protocol used in the GIFT-CF3 study (NCT04618185) to measure GI physiology in addition to MRI measures of lung and liver structure and function. The aim is to identify whether these measures are changed before and after starting ETI.

For the CF participants, to be enrolled in the study they must be homozygous or have at least 1 copy of the Phe508del mutation, which would mean they are eligible for ETI treatment.

The modified MRI protocol, taken from NCT04618185, has been shortened to include scans that are taken over three timepoints. These timepoints are determined around the ingestion of a test meal which has been previously described. Participants will arrive fasted before having a baseline scan. After their first scan they will eat their first standardised high fat meal followed by a second standardised high fat meal around 240 minutes after.

MRI scans to assess GI function will be taken at baseline (fasted), 240 minutes post ingestion of a breakfast meal (T240) and 300 minutes post breakfast (T300). Liver scans will also be taken at baseline and lung scans taken opportunistically at the T240 timepoint. In total, participants will be asked to remain in the MRI scanner for approximately 30 minutes at a time. For comfort, participants will be able to watch multimedia programmes through the use of a specially adapted television while in the scanner.

Participants will also be asked to complete validated gastrointestinal questionnaires throughout the study day and recall their GI symptoms over the previous 2 weeks and complete a 3 day food diary.

The study will be split into two phases. The first will be a pilot phase where 3 children with CF aged 6 to 11 years and 3 healthy age and gender matched controls undergo MRI scanning. These scans will be assessed to determine whether the scan protocol can be completed by the participants and assess the quality of the images obtained. If successful, the trial will progress onto the main phase.

In the main phase, the 12 additional children with CF will be recruited and undergo the above scanning protocol, prior to starting ETI. We will then ask participants to return for a repeat scans approximately 6 months after starting ETI.

ELIGIBILITY:
Inclusion Criteria:

* Children with CF aged 6 to 11 years. Must have at least one copy of the Phe508del mutation.
* Healthy volunteers must have no previous history of gastrointestinal disease.

Exclusion Criteria:

* Healthy volunteers with a history of gastrointestinal disease.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with CF aged 6 to 11 years. Must have at least one copy of the Phe508del mutation. These children would be planned to start receiving ETI as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Delta Small Bowel Water (DeltaSBW) | This a measure of the change in small bowel water between study time points 240 minutes and 300 minutes post first study meal.
  This measurement relates to the postprandial fall in small bowel water content post second study meal. This will be adjusted to body surface area (mL/m2)

SECONDARY OUTCOMES:
Small bowel water content | Will be measured at study timepoints: baseline, 240 minutes and 300 minutes and then area under the curve calculated using the three timepoints (L.min/m2)
  Volume of small bowel water within the small bowel, adjusted to body surface area (mL/m2)
Liver volume | Measured during fasted, baseline MRI scan
  Measurement of total liver volume during fasted baseline scan
Liver elastography | Measured during fasted, baseline MRI scan
  Measurement of liver firmness using MRI elastography
Lung ventilation | Measured at 240 minute time point
  Measured using phase-resolved functional lung (PREFUL) MRI sequence

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Prayle, Principal Investigator — Associate Professor; Alan Smyth, Principal Investigator — Professor of Child Health
Locations (1):
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom